CLINICAL TRIAL: NCT05926167
Title: VALIDATE II Study: Observational Trial Evaluating Elevated Factor VIII Related Labs in Multiple Sclerosis Relapse as a Marker for Incomplete Recovery
Brief Title: Observational Trial Evaluating Elevated Factor VIII Related Labs as a Biomarker for Incomplete Relapse Recovery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dignity Health Medical Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Validate II
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Multiple Sclerosis; Relapse
Keywords: multiple sclerosis relapse biomarker; Factor VIII
MeSH Terms: conditions — Multiple Sclerosis; Recurrence; Hemophilia A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: blood tests drawn days 1, 8, 22 and 90 of the study — Blood tests related to Factor VIII activity that are not a part of standard of care

SUMMARY:
Nine Multiple Sclerosis (MS) patients suffering an acute relapse from the outpatient or inpatient settings will be consented to be followed prospectively for three months post relapse, in an effort to identify markers of incomplete relapse recovery. Factor VIII-related labs will be drawn for three months without influencing standard of care treatment decisions. During this time, patients will be followed with clinical and diagnostic assessments in addition to blood tests including: Expanded Disability Status Scale (EDSS), Multiple Sclerosis Functional Composite (MSFC), recovery surveys, and MRIs of the brain, cervical spine, and thoracic spine with and without contrast. Clinical, imaging, and Factor VIII-related lab data individually or in aggregate will be correlated with relapse presence, severity, and extent of recovery following standard treatment interventions.

DETAILED DESCRIPTION:
The identification of blood tests that detect patients having disability provoking Multiple Sclerosis (MS) relapses in real time could lead to a new era of MS relapse treatment. The cross-talk between inflammatory and coagulation pathways in multiple sclerosis has been recognized on some level for decades. Accidental and anecdotal clinical observations suggest that excessive activation of the intrinsic coagulation pathway, namely with increased Factor VIII activity, occurs with some MS relapses, and that these are the relapses that don't recover with current standard of care treatments, leaving behind permanent disability.

To test this hypothesis that real time abnormally increased levels of Factor VIII activity related labs can identify disabling relapses in real time, nine adult patients with relapsing remitting MS with or without secondary progression will be consented and enrolled in this observational, longitudinal clinical trial. Patients will receive standard of care treatment per the investigator's discretion for their relapse, but will have additional blood tests testing Factor VIII activity, Factor VIII antigen, serum neurofilament among others drawn on days 1, 8, 22 and 90 of the study. The investigator and the patient will not know these lab test results. Patients will also have mris of the brain, cervical spine, and thoracic spine done with and without contrast as soon as possible upon study entry. On Days 1,8,22, and 90, in addition to blood tests, the patient will complete an EDSS and MSFC (that looks at ambulation, hand/arm coordination, and cognitive function, comprised of the 25 foot timed walking tests, with and without any assistive devices if possible), and fill out a recovery survey. Individual blood tests, aggregate blood tests, mri findings, EDSS and MSFC individual and summed scores will be scrutinized and evaluated for the ability to identify a MS relapse and to identify a treatment-resistant MS relapse

ELIGIBILITY:
Inclusion Criteria: Identified by prinicipal investigator as having an acute multiple sclerosis relapse of less than 30 days duration

-

Exclusion Criteria:

Inability to have a MRI

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult relapsing remitting patients with an established or new diagnosis of relapsing remitting multiple sclerosis suffering an acute MS relapse. Patients can be on any disease modifying therapy or on no therapy. Patients who cannot have a MRI, found to have an alternative neurological explanation for their symptoms will be excluded. Patients will be enrolled from a Multiple Sclerosis clinic or from an inpatient hospital setting.
Sampling Method: Probability Sample
Enrollment: 9 (Estimated)
Dates: Start 2023-09-12 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Correlation of Factor VIII activity, Factor VIII with MS relapse | 90 days
Correlation of Factor VIII activity, Factor VIII antigen with MS relapse incomplete recovery | 90 days
Correlation of additional labs with MS relapse or MS relapse incomplete recovery | 90 days
Correlation of MRI findings with MS relapse and MS relapse recovery | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Sabeen B Lulu, MD, Principal Investigator — Dignity Health Medical Foundation